CLINICAL TRIAL: NCT06798363
Title: Efficacy and Safety of Different Initial Doses of Oral Propranolol in the Treatment of Ulcerated Infantile Hemangioma： a Prospective Study
Brief Title: Efficacy and Safety of Different Initial Doses of Oral Propranolol in the Treatment of Ulcerated Infantile Hemangioma
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Yi Ji, Doctor, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RCT20250123
Record Dates: First submitted 2025-01-23; First posted 2025-01-29 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Infantile Hemangioma
Keywords: Infantile hemangioma, ulcer, propranolol
MeSH Terms: conditions — Hemangioma, Capillary; Ulcer | interventions — Propranolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- low dose (Experimental): 1mg/kg/d
  Interventions: Drug: propranolol
- high dose (Active Comparator): 2mg/kg/d
  Interventions: Drug: propranolol

INTERVENTIONS:
Drug: propranolol — different dose

SUMMARY:
The main objective of this study was to determine the efficacy of different doses of propranolol in the treatment of ulcerattion infantile hemangioma (IH).

DETAILED DESCRIPTION:
Infantile hemangioma (IH) is the most common benign tumor in infants, with an estimated prevalence of 4%-5%. Although most IH resolves over time without serious sequelae, a significant proportion can lead to serious complications such as ulcers. Propranolol is considered to be an effective treatment modality for ulceration IH, and there are retrospective studies suggesting that starting treatment at a low dose is safe and effective. However, due to the lack of prospective study, the effectiveness of different doses of propranolol for initiating treatment of ulceration IH is unknown. Therefore, a prospective study of ulceration IHs in Chinese children was conducted to clarify its efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. all patients with ulcer IH;
2. children with ulcer IH treated with propranolol.

Exclusion Criteria:

1) children with ulcer IH who received other therapeutic interventions were excluded; 2) Children whose families refused to participate in the study; 3) patients with contraindications to oral propranolol, such as allergy to propranolol, severe bradycardia and bronchial asthma; 4) children lost to follow-up during oral propranolol treatment; 5) children unable to oral propranolol or continue to oral propranolol due to other reasons.

-

Ages: 1 Month to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2025-04-02 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Time to ulcer healing | 1.5 years
  Time from the start of treatment with propranolol to complete ulcer healing

SECONDARY OUTCOMES:
The resolution of IH at month 6 after treatment | 1.5 years
  complete resolution/complete resolution/partial resolution/no effect/withdrawal from treatment
adverse events | 1.5 years
  The incidence of adverse events in the two groups after oral propranolol at different doses

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital of Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No